CLINICAL TRIAL: NCT05090514
Title: Ready to Read: A School-Based Intervention to Promote Growth Mindset and Reading
Brief Title: Ready to Read: Ready to Read: A School-Based Intervention to Promote Growth Mindset and Reading
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Irene M. Loe, MD, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61892
Record Dates: First submitted 2021-09-28; First posted 2021-10-22 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Reading
Keywords: Reading; Growth Mindset

STUDY DESIGN:
Intervention Model Description: Demonstration project in an underserved, urban school with children randomized to intervention group or wait-list control group.
Who Masked: Outcomes Assessor
Masking Description: The primary outcome, reading achievement, is measured by school personnel who are not aware of the child's study group status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reading and Growth Mindset Intervention Group (Experimental): Parents and students receive a packet of age-appropriate books and educational materials on how to read together/promote reading with their child using growth mindset strategies and where to find other reading materials. Parents also receive 2 weekly text messages with tips and reminders to read with their child daily for 20 minutes over the course of 8 weeks. The messages contain a link to a secure Redcap survey to log days and time spent reading the prior week.
  Interventions: Behavioral: Reading and Growth Mindset
- Wait-list Control Group (Active Comparator): Parents and students receive a packet of age-appropriate books at the same time as the intervention group, but do not receive specialized instruction or reminders to read.
  Interventions: Behavioral: Wait-list Control

INTERVENTIONS:
Behavioral: Reading and Growth Mindset — Parents and students receive a packet of age-appropriate books and educational materials (flyer/handouts, link to educational video) on how to read together/promote reading with their child using growth mindset strategies and where to find other reading materials. Parents also receive 2 weekly text messages with tips and reminders to read with their child daily for 20 minutes over the course of 8 weeks. The messages contain a link to a secure Redcap survey to log days and time spent reading the prior week.
  Arms: Reading and Growth Mindset Intervention Group
Behavioral: Wait-list Control — Parents and students receive a packet of age-appropriate books at the same time as the intervention group, but do not receive specialized instruction or reminders to read or any information on growth mindset and reading.
  Arms: Wait-list Control Group

SUMMARY:
Primary Aim/Objective: To determine if a school-based intervention promoting reading with a growth mindset framework improves student reading achievement in the intervention group compared to a wait-list comparison group of children in kindergarten through 2nd grade.

Secondary Aim/Objective: To determine if students whose parents endorse a fixed mindset with regard to student reading abilities show more improvement post-intervention than parents that endorse growth mindset.

Secondary Aim/Objective: To determine if more parents endorse growth than fixed mindset post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* all children in kindergarten through 2nd grade and their caregivers at the targeted elementary school

Exclusion Criteria:

* Less than kindergarten or above 2nd grade

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Reading Achievement on the Fountas and Pinnell Benchmark Assessment System | Administered at baseline and through intervention completion, an average of 8 weeks
  Change in standardized reading achievement scores collected by the school district to assess reading comprehension, fluency, phonemic awareness.

SECONDARY OUTCOMES:
Change in Parent Growth Mindset as applied to Reading | Administered at baseline and through intervention completion, an average of 8 weeks
  Change in parent growth mindset as assessed by 6 mindset questions based on prior studies on reading abilities in children, assessed on a 6-point Likert scale. Modeled after the classic Growth Mindset of Intelligence questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Irene M Loe, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No